CLINICAL TRIAL: NCT05193162
Title: Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, No. 197 Ruijin Road II, Shanghai 200025, China
Brief Title: Retrospective Study on Microbial Diversity in Paraffin Tissue of Pancreatic Diseases
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, WeiWang, Chief physician, Ruijin Hospital
Other Study IDs: (2021)Clin. Ethics Appr. (257)
Record Dates: First submitted 2021-12-31; First posted 2022-01-14 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Pancreatic Cancer; Pancreatic Disease; Microbial Colonization
Keywords: Pancreatic cancer; Pancreatic Diseases; Microbial Colonization
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Diseases; Communicable Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Collect lesion tissue samples and extract DNA. The lesion tissues were obtained from the paraffin tissues which were made from the surgical specimens for sampling.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Pancreatic ductal adenocarcinoma: According to the relevant information such as clinical features and prognosis, it may continue to be divided into several subgroups.
  Interventions: Other: No any intervention
- Chronic pancreatitis: According to the relevant information such as clinical features and prognosis, it may continue to be divided into several subgroups.
  Interventions: Other: No any intervention
- Pancreatic serous cystadenoma: According to the relevant information such as clinical features and prognosis, it may continue to be divided into several subgroups.
  Interventions: Other: No any intervention
- Pancreatic mucinous cystadenoma: According to the relevant information such as clinical features and prognosis, it may continue to be divided into several subgroups.
  Interventions: Other: No any intervention
- Intraductal papillary mucinous tumor: According to the relevant information such as clinical features and prognosis, it may continue to be divided into several subgroups.
  Interventions: Other: No any intervention
- Pancreatic neuroendocrine tumor: According to the relevant information such as clinical features and prognosis, it may continue to be divided into several subgroups.
  Interventions: Other: No any intervention
- Pancreatic acinar cell carcinoma: According to the relevant information such as clinical features and prognosis, it may continue to be divided into several subgroups.
  Interventions: Other: No any intervention
- Solid pseudopapillary tumor of pancreas: According to the relevant information such as clinical features and prognosis, it may continue to be divided into several subgroups.
  Interventions: Other: No any intervention
- Blank paraffin section
  Interventions: Other: No any intervention

INTERVENTIONS:
Other: No any intervention — have no any intervention
  Other Names: have no any intervention

SUMMARY:
The great harm of pancreatic diseases and the unknown etiology and pathogenesis make it difficult to intervene in most early cases in time. Previous studies by scholars and applicants at home and abroad have shown that the microflora in pancreatic tissue is closely related to chronic pancreatitis and pancreatic cancer. However, the research on the mechanism of microbial diversity in pancreatic tissue and the occurrence and development of various pancreatic diseases has not been reported. Based on the previous research, this subject continues to take various pancreatic diseases as the research object based on the database of pancreatic center and pathology department of Ruijin Hospital Affiliated to Medical College of Shanghai Jiaotong University, To explore the characteristics of microbial flora in pancreas in different pancreatic diseases and its mechanism of influence on disease microenvironment. Select specific microbial flora or targets in the pancreas for various pancreatic diseases, so as to provide new theoretical basis and practical guidance for the early diagnosis and treatment of pancreatic diseases.

DETAILED DESCRIPTION:
AIMS:

To explore the correlation between the characteristics of microbial flora in pancreas and clinical and pathological characteristics of patients with various pancreatic diseases; To clarify the similarities and differences of microbial flora in pancreas in different pancreatic diseases; Select the specific microbial flora or targets in the pancreas for various pancreatic diseases; To provide a new theoretical basis and practical guidance for the early diagnosis, treatment and prognosis of pancreatic diseases.

METHODS:

（1）Patients with various pancreatic diseases operated from January 2005 to June 2022, including but not limited to: pancreatic ductal adenocarcinoma, chronic pancreatitis, pancreatic serous cystadenoma, pancreatic mucinous cystadenoma, intraductal papillary mucinous tumor, pancreatic neuroendocrine tumor, pancreatic acinar cell carcinoma, solid pseudopapillary tumor of pancreas and other pancreatic diseases.

(2) According to the database of Ruijin Hospital, about 30 age and sex matched cases were selected for each pancreatic disease.

(3) All the participants provided written informed consent for participating in the study. If the patient dies, there is an ethical exemption. The collecting procedures have no intervention or impact on treatment measures.

(4)The lesion tissue and adjacent pancreatic tissue were obtained from the paraffin tissue made from the surgical specimens for sampling.

(5)High throughput sequencing was performed according to the instructions of 16S rRNA gene sequencing kit or macro gene detection kit. Anosim (analysis of similarities) statistical method was used for similarity analysis to analyze the correlation between microbiota differences and patients' clinical characteristics (including but not limited to various clinical symptoms, serological indexes, tumor stage, prognosis, and human whole exon sequencing, etc.), pathological type and grade, whether to transfer or not.

(6)According to the instructions of immunohistochemical detection and immunofluorescence detection, the relative abundance and localization of microorganisms in different pancreatic tissues of different pancreatic diseases in different cells (tumor cells, immune cells, normal pancreatic acinar cells, duct cells, etc.) were detected.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 5 years old, ≤ 85 years old;
* After MDT discussion, routine surgery can be performed, and the postoperative pathology is clear as pancreatic cancer and other pancreatic diseases;
* No history of antibiotics for three months before surgery, no history of yogurt containing probiotics
* There is no serious damage to heart, liver and kidney function.

Exclusion Criteria:

* Antibiotics or yogurt containing probiotics history in three months;
* Patients with evidence of sensory or motor neuropathy;
* Those who have a clear cardiovascular disease, severe associated disease or active infection, including known HIV infection;
* Those who have a history of other cancers.

Ages: 5 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male / Female, Age ≥ 5 years old, ≤ 85 years old; - After MDT discussion, routine surgery can be performed, and the postoperative pathology is clear as pancreatic cancer and other pancreatic diseases; - No history of antibiotics for three months before surgery, no history of yogurt containing probiotics - There is no serious damage to heart, liver and kidney function.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
16sRNA and metagenomics | 7/2026
  To obtain intestinal microbial information in patients with pancreatic cancer and other pancreatic diseases, to obtain microbial community structure, evolutionary relationship and information on microbial and environmental correlation in the intestinal environmental samples (weight unit: gram). The patient's microbiological characteristics were correlated with the patient's clinical characteristics and prognosis, so as to obtain the relevant biomarker information.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, Dr., Study Chair — Ruijin Hospital, School of Medicine, Shanghai Jiao Tong University，No. 197 Ruijin Road II
Locations (1):
- Ruijin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided